CLINICAL TRIAL: NCT05916443
Title: Study of the Biology of Colorectal Cancer in Early-onset Patients
Brief Title: Dissecting the Biology of Early-onset Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5527
Record Dates: First submitted 2023-05-08; First posted 2023-06-23 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-04

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Contrarily to late-onset (LO) colorectal cancer (CRC), early-onset (EO) CRC incidence is increasingly growing. Several factors, such as obesity, chronic inflammation, and intestinal dysbiosis, can increase the general risk of CRC. However, little is known about the biology of EO-CRC. To evaluate whether such selective rise in the incidence of EO-CRC patients mirrors a distinct transcriptomic profile, the investigators will first dissect EO-CRC's transcriptomic landscape.

Then, the investigators will investigate the colorectal cancer stem cell (CSC) compartment by in vitro functional assays and RNA-seq analysis. Because our preliminary data indicate an increased aggressiveness of the tumor microenvironment (TME) in EO-CRC,the investigators propose to investigate the CSC niche and the interaction with the TME to dissect the molecular and cellular pathways occurring in EO-CRC.

A cohort of 30 EO-CRC patients (<50 years old) will be enrolled and fully characterized. About 10 EO-CRC-derived CSCs in the form of organoids and spheroids will be generated. Since the relevant differences between CR-CSCs isolated from EO-CRC vs LO-CRC patients are still unknown, the investigators will gain information about their specific features such as clonogenic activity, tumorigenic/invasive capacity, and about differences in the mechanisms regulating their cross-talk with TME components.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 and < 50 years ;
* Written informed consent

Exclusion Criteria:

* Non-availability of informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: National multicenter study, enrolling approximately 30 patients with colorectal cancer, males and females, no pediatric age.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Isolation and characterization of EO-CRC-derived CSCs | 2 years
  Identification of EO-CRC-derived CSCs by cytofluorimetry and immunofluorescence analyses (Percentage of cells positive for CD133, CD24, CD44 and CD44v6 expression).
Identification of obesity-associated adipokines in EO-CRC obese patients | 2 years
  Elisa/Luminex assay evaluation of obesity-associated adipokines concentration
Identification of EO-CRC specific signatures and pathways | 2 years
  RNAseq data analysis of differentially expressed genes in EO-CRC-derived CSCs compared with LO-CRC-derived CSCs.